CLINICAL TRIAL: NCT01698073
Title: Teen Pregnancy Prevention Among Native Youth of the Northern Plains
Brief Title: Effect of a Culturally-based Intervention on Sexual Risky Behavior Among Young American Indian Adolescents
Acronym: COL/AS+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-0241
Record Dates: First submitted 2012-09-25; First posted 2012-10-02 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Teen Pregnancy Prevention
Keywords: Teen pregnancy prevention; American Indian; Group-randomized trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mCOL (Experimental): mCircle of Life is a culturally-based HIV-prevention intervention designed for American Indian and Alaska Native 10-12 year-olds. It includes both online and facilitated material.
  Interventions: Behavioral: mCOL
- AS+ (Active Comparator): After-School Science Plus is a curriculum designed for youth to teach science and literacy using everyday materials. It helps youth see how science is a part of everyday life and provides role models of scientists who come from different backgrounds and ethnicities.
  Interventions: Other: AS+

INTERVENTIONS:
Behavioral: mCOL
  Other Names: mCircle of Life
  Arms: mCOL
Other: AS+
  Other Names: After-School Science Plus
  Arms: AS+

SUMMARY:
Youth who participate in the Circle of Life (COL) program will report less sexual risk taking behavior compared to youth who do not receive the program.

DETAILED DESCRIPTION:
Youth who participate in the Circle of Life (COL) program will report less sexual risk taking behavior and fewer pregnancies compared to youth who do not receive the program.

ELIGIBILITY:
Inclusion Criteria:

* 10-12 years old at baseline
* A member of participating Native Boys and Girls Club
* Signed Parental Consent Form
* Signed Parental Permission Form
* Signed Child Assent Form

Exclusion Criteria:

* None Noted

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 167 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Ever had sexual intercourse | Baseline, 3 months, 1 year
  Ever had sexual intercourse is measured by youth self-reported answers in an online survey to a question on lifetime sexual activity. Specifically, youth are coded "1" if they report having had sex ever before in their lifetimes, "0" otherwise. This question is repeated at each data collection point with youth.

CONTACTS AND LOCATIONS:
Overall Officials: Carol E Kaufman, PhD, Principal Investigator — University of Colorado Anschutz Medical Campus, Centers for American Indian and Alaska Native Health
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Background] Kaufman CE, Litchfield A, Schupman E, Mitchell CM. Circle of Life HIV/AIDS-prevention intervention for American Indian and Alaska Native youth. Am Indian Alsk Native Ment Health Res. 2012;19(1):140-53. doi: 10.5820/aian.1901.2012.140. PMID 22569729
- [Background] Kaufman CE, Whitesell NR, Keane EM, Desserich JA, Giago C, Sam A, Mitchell CM. Effectiveness of Circle of Life, an HIV-preventive intervention for American Indian middle school youths: a group randomized trial in a Northern Plains tribe. Am J Public Health. 2014 Jun;104(6):e106-12. doi: 10.2105/AJPH.2013.301822. Epub 2014 Apr 22. PMID 24754555
- [Derived] Black KJ, Morse B, Tuitt N, Big Crow C, Shangreau C, Kaufman CE. Beyond Content: Cultural Perspectives on Using the Internet to Deliver a Sexual Health Intervention to American Indian Youth. J Prim Prev. 2018 Feb;39(1):59-70. doi: 10.1007/s10935-017-0497-0. PMID 29344773